CLINICAL TRIAL: NCT05771480
Title: A Phase IIIb, Single Arm, Open-label, Multicentre Study of Durvalumab in Combination With Chemotherapy for the First Line Treatment for Patients With Advanced Biliary Tract Cancers (TOURMALINE)
Brief Title: Durvalumab With Chemotherapy as First Line Treatment in Patients With Advanced Biliary Tract Cancers (aBTCs)
Acronym: TOURMALINE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4191C00140; 2022-502043-35 (Registry Identifier: CTIS (EU)); 2022-002527-35 (EudraCT Number)
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Biliary Tract Cancer
Keywords: monoclonal antibodies; PD-L1 antagonist; Durvalumab
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab; Gemcitabine; Cisplatin; gemcitabine-oxaliplatin regimen; Carboplatin; S 1 (combination); Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a single arm study with durvalumab in combination with investigator's choice of 7 different background gemcitabine-based chemotherapy regimens in participants with aBTC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Gemcitabine based chemotherapy (Experimental): Participants will receive durvalumab 1500mg every 3 or 4 weeks, in combination with continuation of all or some of the original background gemcitabine based chemotherapy every 3 or 2 weeks for up to a maximum of 8 cycles of chemotherapy. Durvalumab 1500mg is given as a 60-minute IV infusion in the first cycle (Day 1) and as a 30-minute IV infusion in following cycles.
  Upon completing 8 cycles of background gemcitabine-chemotherapy, or after discontinuing any of the combination chemotherapies due to toxicity before completing 8 cycles, participants are eligible to continue receiving durvalumab 1500 mg IV every 4 weeks either alone or in combination with gemcitabine-based chemotherapy (with the exception of paclitaxel), as per investigator's discretion.
  Interventions: Biological: Durvalumab; Drug: Gemcitabine monotherapy; Drug: Gemcitabine + cisplatin; Drug: Gemcitabine + oxaliplatin; Drug: Gemcitabine + carboplatin; Drug: Gemcitabine + cisplatin + S-1; Drug: Gemcitabine + S-1; Drug: Gemcitabine + cisplatin + albumin-bound paclitaxel

INTERVENTIONS:
Biological: Durvalumab — Participants will receive 1500 mg every 3 weeks, or every 4 weeks (in combination with chemotherapy every 3 weeks, or every 2 weeks, respectively) from cycle 1 to cycle 8 of chemotherapy. Upon completion, participants will receive 1500 mg every 4 weeks (as monotherapy)
  Other Names: Background Gemcitabine-based Chemotherapy Regimen
Drug: Gemcitabine monotherapy — Gemcitabine monotherapy as background gemcitabine-based chemotherapy every 3 weeks (i.e., 8 cycles of durvalumab)
  Other Names: Background Gemcitabine-based Chemotherapy Regimen
Drug: Gemcitabine + cisplatin — Gemcitabine plus cisplatin as background gemcitabine-based chemotherapy every 3 weeks (i.e., 8 cycles of durvalumab) for WHO/ECOG PS 2 participants only
  Other Names: Background Gemcitabine-based Chemotherapy Regimen
Drug: Gemcitabine + oxaliplatin — Gemcitabine + oxaliplatin as background gemcitabine-based chemotherapy every 3 weeks (i.e., 8 cycles of durvalumab)
  Other Names: Background Gemcitabine-based Chemotherapy Regimen
Drug: Gemcitabine + carboplatin — Gemcitabine + carboplatin as background gemcitabine-based chemotherapy every 3 weeks (i.e., 8 cycles of durvalumab)
  Other Names: Background Gemcitabine-based Chemotherapy Regimen
Drug: Gemcitabine + cisplatin + S-1 — Gemcitabine + cisplatin + S-1 as background gemcitabine-based chemotherapy every 2 weeks (i.e, 4 cycles of durvalumab)
  Other Names: Background Gemcitabine-based Chemotherapy Regimen.; This regimen is not allowed for countries in the European Union.
Drug: Gemcitabine + S-1 — Gemcitabine + S-1 as background gemcitabine-based chemotherapy every 3 weeks (i.e., 8 cycles of durvalumab)
  Other Names: Background Gemcitabine-based Chemotherapy Regimen; This regimen is not allowed for countries in the European Union.
Drug: Gemcitabine + cisplatin + albumin-bound paclitaxel — Gemcitabine + cisplatin + albumin-bound paclitaxel as background gemcitabine-based chemotherapy every 3 weeks (i.e., 8 cycles of durvalumab)
  Other Names: Background gemcitabine-based chemotherapy Regimen; This regimen is not allowed for countries in the European Union.

SUMMARY:
A study to assess the safety and efficacy of durvalumab in combination with gemcitabine-based chemotherapy regimens in participants with aBTC.

DETAILED DESCRIPTION:
This study involves assessing the safety and efficacy of durvalumab in combination with different gemcitabine-based chemotherapy regimens as first line therapy for aBTC. The target population of interest in this study is participants with aBTC who are ≥ 18 years of age and above legal age per local regulations with WHO/ECOG PS of 0 to 2 at enrolment and who are not eligible for locoregional therapy. Participants with WHO/ECOG PS 2 will be capped at 20% of the overall treated participant population.

The study consists of 4 periods: screening period (Day-28 to Day -1), treatment period up to 8 cycles of gemcitabine-based chemotherapy regimens with durvalumab, maintenance treatment with durvalumab alone or in combination with gemcitabine-based chemotherapy (with the exception of paclitaxel), and then safety and survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable advanced or metastatic biliary tract carcinoma (BTC) including cholangiocarcinoma (intrahepatic or extrahepatic), gallbladder carcinoma, and ampulla of Vater (AoV) carcinoma
* Participants with unresectable or metastatic BTC
* A World Health Organisation Eastern Cooperative Oncology Group Performance Status (WHO/ECOG PS) of 0 to 2
* At least one lesion that qualifies as a Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) target lesion at baseline
* Adequate organ and bone marrow function
* Body weight of > 30 kg
* Negative pregnancy test (serum) for women of childbearing potential
* Female participants must be one year post-menopausal (amenorrhoeic for 12 months without an alternative medical cause)
* Male and female participants and their partners must be surgically sterile or on their chosen method of birth control as per the protocol.

Exclusion Criteria:

* Any evidence of diseases such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diseases, active infection, active interstitial lung disease/pneumonitis, serious chronic gastrointestinal conditions associated with diarrhoea, psychiatric illness/social situations, history of uncontrolled or symptomatic cardiac disease, and history of allogenic organ transplant
* Active or prior documented autoimmune or inflammatory disorders
* History of another primary malignancy, except for malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study intervention
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Known to have tested positive for human immunodeficiency virus [HIV] (positive HIV 1/2 antibodies) or active tuberculosis infection
* Participants co-infected with Hepatitis B virus (HBV) and Hepatitis C virus (HCV) or co-infected with HBV and Hepatitis D virus (HDV)
* Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade > 1) caused by previous anticancer therapy
* Central nervous system metastases requiring treatment or history of spinal cord compression
* Known allergy or hypersensitivity to any of the study intervention or any of the study intervention excipients.
* Any concurrent chemotherapy, other than the one allowed in the study, investigational medicinal product (IMP), biologic, or hormonal therapy for cancer treatment
* Palliative radiotherapy with a limited field of radiation within 2 weeks of the first dose of study intervention, or radiotherapy with a wide field of radiation or radiotherapy affecting more than 30% of the bone marrow within 4 weeks before the first dose of study intervention
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention
* Major surgical procedure within 28 days prior to the first dose of IMP
* Prior exposure to immune-mediated therapy excluding therapeutic anticancer vaccines
* Receipt of the last dose of anticancer therapy within 28 days prior to the first dose of IMP

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Grade 3 or 4 possibly related adverse event (PRAE) | Within 6 months after the initiation of Investigational Medicinal Product (IMP)
  PRAE is defined as an AE which has been assessed by the investigator to be possibly related to IMP.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of the first dose of IMP until death due to any cause [approx. upto 33 months]
  OS is defined as the time from the date of the first dose of IMP until death due to any cause.
Objective Response Rate (ORR) | From the date of first dose of IMP until progression, or the last evaluable assessment in the absence of progression [assessed up to 33 months]
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, as determined by the investigator at local site per RECIST 1.1.
Progression-Free Survival (PFS) | From the date of the first dose of IMP until until the date of objective PD or death [approx. up to 33 months]
  PFS is defined as the time from the first dose of IMP until the date of disease progression (PD) or death due to any cause.
Disease Control Rate (DCR) | Week 24 and Week 32
  DCR is defined as the % of participants who have a best objective response of complete response or partial response (by week 24 or 32), or who have stable disease for 24 or 32 weeks.
Duration of Response (DOR) | From the date of first documented response until the first date of documented progression or death in the absence of disease progression [approx. up to 33 months]
  DOR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Duration of Treatment (DOT) | From date of start of IMP, until 27 days after last dose of IMP or date of death [approx. up to 33 months]
  DOT is defined as time on study intervention.
Number of participants with AEs, including PRAEs, adverse events of special interest (AESIs), immune-mediated adverse events (imAEs) and serious adverse events (SAEs) | From the date of first dose of IMP until long-term follow-up i.e. until 90 days following discontinuation of the last dose of IMP [approx. up to 33 months]
  To assess the safety and tolerability profile of durvalumab combined with background gemcitabine-based chemotherapy
Number of participants with IRRs and hypersensitivity/anaphylactic reactions | From the date of first dose of IMP until 90 days following discontinuation of the last dose of IMP [approx. up to 33 months]
  To assess the safety and tolerability profile of durvalumab combined with background gemcitabine-based chemotherapy
European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ C-30) | From date of first dose of IMP, until the date of the first clinically meaningful deterioration [approx. up to 33 months]
  To assess disease and treatment related symptoms and HRQoL. EORTC QLQ-C30 consists of 30 items and measures symptoms, functioning, and global health status/QoL for all cancer types. Questions are grouped into 5 multi-item functional scales (physical, role, emotional, cognitive, and social), 3 multi-item symptom scales (fatigue, pain, and nausea/vomiting), a 2-item global QoL scale, 5 single items assessing additional symptoms commonly reported by cancer participants (dyspnoea, loss of appetite, insomnia, constipation, and diarrhoea), and one item on the financial impact of the disease. The EORTC QLQ-C30 is a valid and reliable PRO instrument in this participant population
EORTC QLQ-BIL21 Score | From date of first dose of IMP, until the date of the first clinically meaningful deterioration [approx. up to 33 months]
  To assess disease- and treatment related symptoms and HRQoL. The EORTC QLQ-BIL21 is a disease-specific (cholangiocarcinoma and cancer of the gallbladder) questionnaire. It consists of 21 items including one question each for side effects, equipment issues, and weight loss, as well as 5 scales (eating symptoms, jaundice symptoms, tiredness, pain, and anxiety). A higher score indicates greater difficulties. The EORTC QLQ-BIL21 is a valid and reliable PRO instrument in this participant population.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (4):
  - Research Site, Mobile, Alabama
  - Research Site, Orange, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Portland, Oregon
- France (4):
  - Research Site, Clichy
  - Research Site, Dijon
  - Research Site, Montpellier
  - Research Site, Villejuif
- Germany (2):
  - Research Site, Chemnitz
  - Research Site, Hanover
- Italy (5):
  - Research Site, Castelfranco Veneto
  - Research Site, Foggia
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Rozzano
- Japan (9):
  - Research Site, Chūōku
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kyoto
  - Research Site, Osaka
  - Research Site, Sendai
  - Research Site, Ube
  - Research Site, Wakayama
  - Research Site, Yokohama
- Research Site, Singapore, Singapore
- Research Site, Seoul, South Korea
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home